CLINICAL TRIAL: NCT03582046
Title: Targeting Abdominal Perfusion Pressure in Septic Shock (The MAP APP Study)
Brief Title: Targeting Abdominal Perfusion Pressure in Septic Shock
Acronym: MAP-APP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of Enrollment
Sponsor: Potrero Medical (Industry)
Collaborators: Emory University (Other); University of Arkansas (Other); Central Arkansas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRD-06-2615
Record Dates: First submitted 2018-06-27; First posted 2018-07-10 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Acute Kidney Injury; Septic Shock; Resuscitations
MeSH Terms: conditions — Acute Kidney Injury; Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Monitoring Group (No Intervention): Patients that sustain intra-abdominal pressure of < 8 mmHg for 48 hours from sepsis diagnosis. Patients will be monitored and given sepsis standard of care.
- Mean Arterial Pressure (MAP) Group (Active Comparator): Patients with elevated intra-abdominal pressure of ≥ 8 mmHg for 48 hours from sepsis diagnosis.
  Interventions: Device: Mean Arterial Pressure (MAP)
- Abdominal Perfusion Pressure (APP) Group (Experimental): Patients with elevated intra-abdominal pressure of ≥ 8 mmHg for 48 hours from sepsis diagnosis.
  Interventions: Device: Abdominal Perfusion Pressure (APP)

INTERVENTIONS:
Device: Abdominal Perfusion Pressure (APP) — Intra-abdominal Pressure (IAP) actively measured and recorded every four hours, and mean arterial pressure (MAP) adjusted to maintain abdominal perfusion pressure (APP) levels ≥ 60 mmHg.
  Other Names: Intra-Abdominal Pressure (IAP)
  Arms: Abdominal Perfusion Pressure (APP) Group
Device: Mean Arterial Pressure (MAP) — Intra-abdominal Pressure (IAP) recorded passively in device, but not measured or reviewed by physician. Patient will be treated with sepsis standard of care, maintaining mean arterial pressure (MAP) of ≥ 65 mmHg.
  Arms: Mean Arterial Pressure (MAP) Group

SUMMARY:
A randomized control trial among patients with septic shock, studying the incidence, progression and recovery of AKI.

DETAILED DESCRIPTION:
Intra-abdominal pressure (IAP) has proven to be an important physiologic parameter in critically ill patients, and elevated IAP can lead to intra-abdominal hypertension (IAH). Literature suggests that IAH is common in patients with septic shock and that there is an association between the presence of IAH and acute kidney injury (AKI) in this group. Mean arterial pressure (MAP) and IAP together help determine the abdominal perfusion pressure (APP) of organs and tissues within the abdominal cavity. Current clinical guidelines for septic shock encourage targeting MAP of 65-70 mmHg with the use of vasopressors after volume resuscitation. However, it remains unclear if hemodynamic support targeting APP: (a) reduces development of acute kidney injury (AKI), (b) decreases progression of AKI, or (c) improves renal recovery rate compared to standard care for severe septic shock patients. A novel Foley catheter and monitoring device, the Accuryn Monitoring System, is capable of detecting physiologic changes in temperature, urine output (UO) and intra-abdominal pressure (IAP). These data streams are captured continuously by a device that is minimally invasive and at a high frequency which, in combination with MAP, allow for a simple calculation of abdominal perfusion pressure (APP). The purpose of this study is to assess kidney function and recovery in septic shock patients and elevated IAP when targeting treatment to maintain APP ≥ 60 mmHg as compared to standard of care targeting MAP of 65-70 mmHg.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (age ≥ 18)
2. Septic shock - identified as early as possible as evidenced by:

   1. Clinical diagnosis of sepsis defined as documented or suspected infection with the use of antibiotic administration OR
   2. Meets qSOFA (Quick Sequential Organ Failure Assessment) Criteria per the Sepsis-3 definitions:

   i. Respiratory rate ≥ 22/min ii. Altered mentation iii. Systolic blood pressure ≤ 100 mmHg AND c. Shock dependent on vasopressor therapy following initial 12-hour Resuscitation Period refractory to further volume expansion as assessed by clinical treatment team; this may be supported by either: i. Lack of blood pressure response following fluid bolus or passive leg raise ii. Hemodynamic data as available (e.g. PPV [positive pressure ventilation], SVV [stroke volume variation], echo, PAOP [pulmonary artery occlusion pressure], right-heart catheterization, etc.)
3. Indication for a urinary bladder catheter (or one currently in place)
4. Indication for an arterial line (or one currently in place at any site)

FOR MONITORING PHASE OF STUDY (MONITORING GROUP)

1. All of the above criteria for the Resuscitation and Observational Periods of the study
2. Intra-abdominal pressure < 8 mmHg

FOR INTERVENTION PHASE OF STUDY (APP VS MAP GROUPS)

1. All of the above criteria for the Resuscitation and Observational Periods of the study
2. Intra-abdominal pressure ≥ 8 mmHg

Exclusion Criteria:

1. Inability to receive a urinary bladder catheter
2. Chronic suprapubic catheter in place
3. Cirrhosis/end stage liver disease, including Child-Pugh class C
4. Severe AKI [acute kidney injury] as defined by life-threatening electrolyte, acidemia, or other indication for imminent emergent dialysis needs within 12 hours of hospital admission
5. Evidence of chronic renal failure stage 5 (including serum creatinine values consistent with CKD 5 [chronic kidney disease, stage 5] or dialysis dependence) in 12-months prior to enrollment
6. Active gastrointestinal bleed likely causing/contributing to the hemodynamic instability
7. Acute intra-abdominal trauma (including intraabdominal surgery within the prior 30 days)
8. Acute pancreatitis with no established source of infection
9. Treating physician deems aggressive care is unsuitable, or has decided to de-escalate care [Do Not Resuscitate (DNR) patients receiving standard care are still eligible]
10. In the opinion of the treating attending physician the patient is unsuitable for the study for any legitimate reason including lack of equipoise, anticipated imminent significant deterioration, anticipated imminent recovery, incarceration, pre-existing medical or psychiatric condition that treating attending physician deems not appropriate for study, or interfering medications
11. Known previous or concurrent enrollment in a treatment clinical trial that, in the opinion of the investigator, might interfere with the objectives/endpoints of this clinical trial
12. Known contraindication to bladder pressure measurement
13. Known pregnancy
14. Suspected or known increased intracranial pressure requiring active neurosurgical consultation
15. Cardiogenic shock requiring extracorporeal support
16. Any requirement for chest compressions prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
Study kidney function by controlling MAP targets to maintain APP levels, in critically ill patients with septic shock and elevated IAP. | 90 days
  To study kidney function and recovery in patients with septic shock and elevated IAP as measured by timed creatinine clearance on calendar days 1-7 when targeting treatment to maintain APP ≥ 60 mmHg with a variable MAP target as compared to standard of care with a fixed MAP target. Creatinine clearance on calendar day 7 post-intervention or on day of ICU discharge, whichever is earliest, is the primary endpoint. Post hospital stay, subjects will have 30 day and 90 day follow up to check subject health status.

SECONDARY OUTCOMES:
Study AKI by controlling MAP targets to maintain APP levels, in patients with IAH treated with standard of care versus patients with septic shock without IAH. | 90 days
  To study the incidence, progression and recovery of AKI as well as patient-centered outcomes among patients with IAH treated by APP target versus standard of care. To study renal injury and recovery and patient-centered outcomes among septic shock patients without IAH.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Connor, MD, Principal Investigator — Emory University School of Medicine, (404) 616-0184 michael.connor@emory.edu; Luis Juncos, MD, Principal Investigator — CAVHS, Little Rock, AR 72205 (501) 257-1000 luis.juncos@va.gov; Nithin Karakala, MD, Principal Investigator — University of Arkansas Medical Center, Little Rock, AR NKarakala@uams.edu
Locations (3):
- United States (3):
  - Central Arkansas Veterans Healthcare System, Little Rock, Arkansas
  - University of Arkansas Medical Center, Little Rock, Arkansas
  - Grady Memorial Hospital, Atlanta, Georgia